CLINICAL TRIAL: NCT02028143
Title: ICE: Intracardiac Ultrasound Within the Left Atrium During Radiofrequency Ablation of Nonvalvular Atrial Fibrillation
Acronym: ICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gregory Jones (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Gregory Jones, Gregory Jones, MD, FACC, Wellmont CVA Heart Institute
Organization: Wellmont CVA Heart Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICE
Record Dates: First submitted 2013-12-31; First posted 2014-01-07 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study arm (Experimental): The study arm group will have the ICE catheter placed through one of two existing 8F sheaths already in the left atrium. The ICE catheter will be exchanged in the sheath utilizing the lasso multipolar mapping catheter during left pulmonary vein ablation lines. During exchange, suction and irrigation techniques will be utilized to avoid any air or thrombus embolization. All patients will have standard anticoagulation during the procedure with heparin infusion adjusted to an activated clotting time (ACT) of 350-400. The left sided ICE catheter will be adjusted to visualize left sided structures, ablation tip and tissue interface, and adjacent noncardiac structures such as the esophagus during radiofrequency ablation of the left pulmonary vein system.
  Interventions: Device: Biosense Webster irrigated tip catheter; Procedure: ICE catheter placed through one of two existing 8F sheaths
- Control arm (Active Comparator): The control arm group will receive standard pulmonary vein isolation (PVI) procedure utilizing intracardiac guided ultrasound (ICE) placed within the right atrium via the femoral vein.
  Interventions: Device: Biosense Webster irrigated tip catheter; Procedure: Pulmonary vein isolation

INTERVENTIONS:
Device: Biosense Webster irrigated tip catheter — The second group (study group) will have the ICE catheter placed through one of two existing 8F sheaths already in the left atrium. The ICE catheter will be exchanged in the sheath utilizing the lasso multipolar mapping catheter during left pulmonary vein ablation lines. During exchange, suction and irrigation techniques will be utilized to avoid any air or thrombus embolization. All patients will have standard anticoagulation during the procedure with heparin infusion adjusted to an activated clotting time (ACT) of 350-400. The left sided ICE catheter will be adjusted to visualize left sided structures, ablation tip and tissue interface, and adjacent noncardiac structures such as the esophagus during radiofrequency ablation of the left pulmonary vein system.
  Other Names: 3.5mm Biosense Webster irrigated tip catheter.
  Arms: Study arm
Device: Biosense Webster irrigated tip catheter — Group 1 will receive standard pulmonary vein isolation (PVI) procedure utilizing intracardiac guided ultrasound (ICE) placed within the right atrium via the femoral vein.
  Other Names: 3.5mm Biosense Webster irrigated tip catheter.
  Arms: Control arm
Procedure: Pulmonary vein isolation
  Arms: Control arm
Procedure: ICE catheter placed through one of two existing 8F sheaths
  Arms: Study arm

SUMMARY:
Imaging Real Time within the Left atrial chamber Enhances safety and efficacy of Radiofrequency Ablation of Atrial Fibrillation

DETAILED DESCRIPTION:
Atrial fibrillation is the most common rhythm disturbance affecting the human population.

1. Its prevalence increases with age and can be found in >8% of humans over the age of eighty;
2. Radiofrequency ablation for drug refractory nonvalvular atrial fibrillation has become a common therapy available to patients. It has been shown to be both efficacious and cost effective;
3. The standard approach to atrial fibrillation involves electrical isolation of the pulmonary veins (PVI) from the rest of the atrium chamber. This involves moving a 3.5mm tip ablation catheter point to point around the PV structures until an encircling ablation line is formed. This can be made difficult by not knowing if the tip is in good contact with the atrial tissue. In addition the esophagus is a posterior lying structure and injury to the esophagus by ablating the overlying tissue has been reported, at times fatal;
4. Currently, intracardiac imaging of the left atrium has FDA approval in the right atrial chamber. This leads to difficulty in visualizing tip tissue interface, and important left sided structures such as carina, ligaments, and esophagus. By placing the tip of the ICE catheter in the left atrium, enhanced visualization of the tip tissue interface may lead to more effective ablation points, fewer needed ablation points, and enhanced safety by avoiding placement over adjacent noncardiac structures.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Recommended for radiofrequency ablation of nonvalvular atrial fibrillation

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
number of lesions requiring ablation to obtain Electrical Isolation PV System | during procedure
  to assess the number of lesions requiring ablation to obtain Electrical Isolation PV system

SECONDARY OUTCOMES:
to assess number of lesions to obtain Electrical Isolation PV system | during procedure
  Evaluate the time required to obtain electrical isolation of PV system

OTHER OUTCOMES:
Safety-Cardiac perforation, emboli, fistula formation | during procedure
  evaluate the use of ultrasound catheter for adverse events such as cardiac perforation, emboli or fistula formation

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Jones, MD, Principal Investigator — Wellmont CVA Heart Institute
Locations (1):
- Wellmont CVA Heart Institute, Kingsport, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No